CLINICAL TRIAL: NCT06435156
Title: A Phase 2 Double-blind Randomised Controlled Trial Studying the Effect of Sotagliflozin Versus Placebo in Individuals With Heart Failure and Type 1 Diabetes.
Brief Title: Sotagliflozin in Patients With Heart Failure Symptoms and Type 1 Diabetes
Acronym: SOPHIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Lexicon Pharmaceuticals (Industry); Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Ify Mordi, MD, Clinical Senior Lecturer and Honorary Consultant Cardiologist, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-50-23; 3-SRA-2023-1376-M-B (Other Grant/Funding Number: Juvenile Diabetes Research Foundation); 1007807 (Other: IRAS)
Record Dates: First submitted 2024-05-16; First posted 2024-05-30 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-02

CONDITIONS: Type 1 Diabetes; Heart Failure
Keywords: Type 1 Diabetes; heart failure; Sodium-glucose Cotransporter-2 (SGLT2) Inhibitors; sotagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Heart Failure | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sotagliflozin (Experimental): Sotagliflozin oral tablet, 200mg once per day for 16 weeks.
  Interventions: Drug: Sotagliflozin
- Placebo (Placebo Comparator): Placebo oral tablet, 200mg once per day for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sotagliflozin — Sodium-glucose Co-transporter inhibitor
  Arms: Sotagliflozin
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
People with type 1 diabetes sometimes develop heart failure which can cause symptoms like breathlessness, tiredness or ankle swelling, reduced quality of life and lead to being admitted to hospital or suffering potential fatal consequences. This trial is investigating if a tablet called sotagliflozin, can improve quality of life in people with type 1 diabetes and heart failure. In addition, this trial will also assess the safety and tolerability of sotagliflozin in this population.

In previous trials that included people with type 2 diabetes and heart failure sotagliflozin was shown to improve patients' symptoms of heart failure, quality of life and reduce the chance of people with heart failure being admitted to hospital or dying. However, people with type 1 diabetes and heart failure were not included in these trials meaning that it is not known if these benefits also apply to this population.

This trial aims to recruit 320 people with type 1 diabetes and heart failure symptoms in multiple sites in the United Kingdom (UK). This trial will compare the health and quality of life of participants who take sotagliflozin tablets with participants who take placebo tablets, which is a dummy tablet that looks the same as sotagliflozin. Participants will be randomly allocated to one of two groups (i.e. one taking sotagliflozin and the other the placebo) and both the medical team and participants will not know in which group each participant is until the end of the study. Participants will be in the trial for approximately 6 months and will be given sotagliflozin or placebo tablets to take 1 per day for 4 months. The trial is expected to run for a total of 26 months.

DETAILED DESCRIPTION:
BACKGROUND Intensive insulin therapy designed to near-normalize glucose levels in people with type 1 diabetes significantly reduces an individual's risk of long-term micro- and macrovascular complications. Unfortunately, glycaemic targets are not achieved by the majority of people with type 1 diabetes and as such overall life expectancy remains reduced compared to those without type 1 diabetes. Cardiovascular disease remains a major cause of morbidity and mortality in type 1 diabetes. There is growing recognition that heart failure (HF) is an increasing problem in type 1 diabetes. Diabetes itself is an independent risk factor for HF, causing structural and functional cardiac changes that predispose to HF (known as diabetic cardiomyopathy). HF is the end result of many cardiovascular diseases such as hypertension and myocardial infarction, and improved treatments for these conditions and changing demographic trends mean that many more people are surviving longer and developing HF.

HF has a substantial healthcare burden. In the United States (US) and Europe, the prevalence of HF in the general population is around 1-2% - around 6 million adults in the US are estimated to be living with HF currently. In 2014 in the US there were ~1.1 million emergency department visits, 980 000 hospitalizations, and 84 000 deaths with HF as the primary cause, with an estimated cost of ~$11.3 billion (~$11,500/per patient for each hospitalisation). Despite advances in management of HF over the past 30 years, the incidence of mortality and HF hospitalisation in recent HF clinical trials remained high at ~20-30% over 2 years.

The burden of HF in type 1 diabetes is less well characterised compared to HF in those with type 2 diabetes (and individuals without diabetes), however the data still indicate the substantial nature of this growing problem. One of the largest epidemiological studies was a Scottish national data study of 3.25 million individuals >30 years old, where the crude incidence of HF hospitalisation was over twice that of the population without diabetes. While the crude incidence was less than in type 2 diabetes, type 1 diabetes patients were on average 20 years younger. Despite their younger age, 30-day mortality following HF hospitalisation was higher in individuals with type 1 diabetes after adjustment for age, sex and socioeconomic status, indicating that outcomes are worse in HF patients with type 1 diabetes compared to those with either type 2 diabetes or without diabetes. Data from Scandinavia supports this finding and suggests that the risk of both incident HF and cardiovascular mortality was higher for individuals with type 1 diabetes compared to type 2 diabetes after adjustment for age. The overall prevalence of HF in this study at baseline was 3.1% - extrapolated to the US this would equate to 57,000 of the 1.9 million individuals with type 1 diabetes. A recent meta-analysis of all available data suggested that the incidence of HF was 3.1 times higher in individuals with type 1 diabetes compared to controls (typically the general population). Assuming a 5% incidence of HF hospitalisation/year, HF hospitalizations cost the US healthcare system ~$29 million per year. In summary, these data suggest that not only is HF a significant problem in individuals with type 1 diabetes, but there is evidence of an outcome disparity compared to individuals with type 2 diabetes or those without diabetes.

Although there are some differences (e.g. presentation at a younger age), the pathophysiology of HF in type 1 diabetes is similar to type 2 diabetes. Risk factors are similar (e.g. glycaemic control, coronary artery disease and hypertension), leading to inflammation, endothelial dysfunction, fibrosis, and subsequent diastolic and systolic dysfunction. Given the pathophysiological similarities, there is little to suggest that HF therapies that have shown benefit in individuals with type 2 diabetes (or individuals without diabetes) would not also be efficacious in type 1 diabetes. In all current HF guidelines mainstay HF treatments (renin-angiotensin system blockers, beta-blockers, and mineralocorticoid receptor antagonists) are recommended for all patients with HF regardless of diabetes status.

Sodium-glucose co-transporter inhibitors (SGLTi) were initially developed as oral add-on treatments for glycaemic control in type 2 diabetes. A consistent finding in large cardiovascular outcome trials was a significant ~30% risk reduction in hospitalisation for HF, as well as overall reductions in cardiovascular mortality. Subsequently, SGLTi in addition to guideline-directed HF therapy have been studied in HF patients either with type 2 diabetes or without diabetes and have again shown a consistent benefit compared to placebo, with significant reductions in mortality and HF hospitalisation irrespective of cardiac function left ventricular ejection fraction (LVEF) at baseline without any concerning safety signals. SGLTi also improve HF-related quality of life (QoL) and renal outcomes. This has led to the inclusion of SGLTi in the most recent HF treatment guidelines as a cornerstone of therapy in addition to established pharmacological agents (e.g., renin-angiotensin system inhibitors, beta-blockers and mineralocorticoid receptor antagonists). However, there is one key issue - individuals with type 1 diabetes have been excluded from these HF trials, in part due to concerns around safety. At present there is no evidence to support the use of these life-saving therapies in this population that already has worse outcomes than other groups with HF.

In adult type 1 diabetes, Phase III trials with dapagliflozin, empagliflozin and sotagliflozin have been completed, collectively showing modest benefits of SGLT inhibition in terms of Haemoglobin A1c (HbA1c) reduction, increased time in range, reduced body weight and total insulin dose. However, SGLTi use in type 1 diabetes was also associated with an increased risk of diabetic ketoacidosis (DKA), which has limited their more widespread use in type 1 diabetes.

Sotagliflozin is a dual SGLT1 and 2 inhibitor that is currently approved in the United Kingdom for use in individuals with type 1 diabetes with a body mass index (BMI) of ≥27kg/m2 and taking insulin doses of at least 0.5 units/kg of body weight in patients with inadequate glycaemic control. As with selective SGLT2i, sotagliflozin also improves HF-related outcomes. The key evidence for this comes from two clinical trials. In the Sotagliflozin in Patients with Diabetes and Chronic Kidney Disease (SCORED) trial including 10,584 patients with type 2 diabetes, chronic kidney disease and cardiovascular risk factors, sotagliflozin caused a 26% relative risk reduction in the primary endpoint of cardiovascular death, HF hospitalisation or urgent HF visit compared to placebo. There was also a 33% relative risk reduction in HF hospitalisation or urgent HF visits, figures consistent with other SGLT2i trials.

The second key trial was the Sotagliflozin in Patients with Diabetes and Recent Worsening Heart Failure (SOLOIST-WHF) trial. In this trial 1,222 patients with type 2 diabetes and a recent HF hospitalisation were randomised to sotagliflozin 200mg once daily (with uptitration to 400mg once daily) or placebo. Patients were included regardless of left ventricular ejection fraction (LVEF) at baseline. The median follow-up duration was 9 months.

Sotagliflozin caused a 33% relative risk reduction in the primary outcome of cardiovascular death, HF hospitalisation or urgent HF visit, with a 36% reduction in HF hospitalisation or urgent HF visits that met statistical significance. Sotagliflozin also significantly improved QoL at 4 months measured using the Kansas City Cardiomyopathy Questionnaire (KCCQ). Rates of serious adverse events (SAEs) leading to study drug withdrawal were similar in both sotagliflozin and placebo groups, though severe hypoglycaemia was more common with sotagliflozin than placebo (9 individuals vs. 2). There was no significant increase in incidence of DKA with sotagliflozin compared to placebo (2 vs. 4). Taken together, these two trials confirm the benefit of sotagliflozin on HF related outcomes, consistent with selective SGLT2i. Again, individuals with type 1 diabetes were excluded from both of these trials.

In summary, there is significant HF related morbidity and mortality in type 1 diabetes, and outcomes are worse than in HF patients with type 2 diabetes or without diabetes. Oral sotagliflozin 200mg daily is licensed for improving glycaemic control in type 1 diabetes in the UK. Although sotagliflozin improves HF related outcomes and QoL in patients with type 2 diabetes and patients with HF who do not have diabetes, studies are needed to determine whether these benefits might extend to patients with type 1 diabetes and heart failure.

RATIONALE As outlined above, HF is a significant problem in type 1 diabetes, with an estimated prevalence of 3-5%. Outcomes for individuals with type 1 diabetes and HF are worse than in those with type 2 diabetes or without diabetes, with increased mortality and hospitalisation rates. Critically, patients with type 1 diabetes have been excluded from pivotal trials of the latest advance in HF treatment (SGLT2i), potentially exacerbating these outcome disparities further.

The proposed trial will be the first to provide data on the efficacy and safety of sotagliflozin, in patients with type 1 diabetes and HF (regardless of LVEF). If a beneficial signal is found, this would provide strong support for extending the use of sotagliflozin in this group of patients with type 1 diabetes and adoption into clinical guidelines. A multi-centre, double-blind, randomised controlled trial to provide the strongest level of evidence for previous findings of the researchers will be conducted. Importantly, by choosing QoL measured using the KCCQ as the primary endpoint, an outcome that not only correlates strongly with mortality and hospitalisation but is also accepted by the US Food and Drug Administration (FDA) as a valid endpoint for regulatory approval has been selected. The KCCQ is a 23- item self-administered questionnaire that measures the patient's perception of their health status, including HF symptoms, impact on physical and social function, and how their HF impacts their QOL within the preceding 2 weeks. Improvements in KCCQ score map very well to reductions in mortality and hospitalisation and SGLT2i have consistently improved KCCQ scores. A 5-point increase in KCCQ score is traditionally considered clinically meaningful and is associated with a 7% reduction in mortality and HF hospitalisation. Given the prohibitive size of trial that would be required to demonstrate an improvement in mortality or HF hospitalizations with sotagliflozin in type 1 diabetes, the KCCQ represents an ideal endpoint for the trial. The proposed trial has the potential to be a high-impact, practice-changing trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to <85 years.
* Type 1 diabetes.
* Insulin dose ≥0.5 units/kg body weight at screening or body mass index (BMI) ≥25kg/m2 at screening
* Using continuous glucose monitor at screening or willing to use one for the duration of the trial.
* Diagnosis of heart failure (HF) regardless of left ventricular ejection fraction (LVEF), defined as one or more of the following:

Previous HF hospitalisation where HF was documented as the primary cause of hospitalisation and there was a requirement for loop diuretics

OR

Impaired left ventricular (LV) function (i.e. LVEF <50% by any imaging modality) at any time

OR

Preserved LV systolic function (LVEF ≥50%) with left atrial enlargement (2-dimensional echocardiographic measurement of left atrial width ≥3.8cm or left atrial length ≥5.0 cm or left atrial area ≥20cm2 or left atrial volume index >29 ml/m2) within the last 24 months.

OR

Preserved LV systolic function (LVEF ≥50%) with left ventricular hypertrophy (2-dimensional echocardiographic measurement of end-diastolic interventricular septal diameter ≥1.2cm or end-diastolic left ventricular posterior wall diameter ≥1.2cm) within the last 24 months.

OR

Preserved LV systolic function (LVEF ≥50%) with echocardiographic diastolic dysfunction (septal e' <7cm/sec or lateral e' <10cm/sec or average E/e' ≥15) within the last 24 months.

* New York Heart Association Class II-IV at screening.
* Elevated N-terminal pro-B-type natriuretic peptide (≥250 ng/L for those in sinus rhythm, ≥400 ng/L if in atrial fibrillation) or B-type natriuretic peptide (≥75 ng/L for those in sinus rhythm, ≥100 ng/L if in atrial fibrillation) within 12 months of screening.
* Kansas City Cardiomyopathy clinical summary score <85 at screening.

Exclusion Criteria:

* Cardiac surgery (coronary artery bypass graft or valve replacement), type 1 myocardial infarction, implantation of cardiac device (including biventricular pacemaker) or cardiac mechanical support implantation within 1 month of screening, or between screening and randomisation, or planned during the trial.
* End-stage heart failure requiring left ventricular assist devices, intra-aortic balloon pump, or any type of mechanical support at the time of randomisation.
* Documented primary severe valvular heart disease, amyloidosis or hypertrophic cardiomyopathy as principal cause of heart failure as judged by the local investigator.
* Respiratory disease thought to be the primary cause of dyspnoea as assessed by the local investigator.
* Chronic kidney disease with estimated glomerular filtration rate <25ml/min/1.73m2 at screening.
* Moderate or severe hepatic impairment (e.g. Child-Pugh B and C) at screening as judged by the local investigator.
* Use of sotagliflozin or any sodium-glucose co-transporter-2 inhibitors (SGLT2i) within 1 month of screening or between screening and randomisation.
* Previous hypersensitivity/intolerance to SGLT2i.
* Presence of malignancy with expected life expectancy <1 year at screening.
* Severe hypoglycaemia (hospitalisation for hypoglycaemia or episode requiring external assistance to treat) within 1 month prior to screening or between screening and randomisation.
* One episode of diabetic ketoacidosis or nonketotic hyperosmolar state within 1 month of screening or between screening and randomisation, or ≥2 diabetic ketoacidosis or nonketotic hyperosmolar state events within 6 months of screening.
* Pregnant or lactating women.
* Women of childbearing age or male partners of women of childbearing age and not practicing an acceptable method of birth control
* On a ketogenic diet.
* Unwilling/unable to share glucose and ketone monitoring data.
* Unwilling to wear continuous glucose monitoring during the trial.
* Use of any investigational drugs within five times of the elimination half-life after the last dose or within 30 days, whichever is longer. Current enrolment in non-interventional, observational studies will be allowed.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire (KCCQ) clinical summary score | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on quality of life (QoL).
  KCCQ clinical summary score (no unit, ranges from 0 to 100 with higher scores reflecting better health status).

SECONDARY OUTCOMES:
Change in KCCQ clinical summary score | From baseline to week 4
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on QoL.
  KCCQ clinical summary score (no unit, ranges from 0 to 100 with higher scores reflecting better health status).
Change in KCCQ overall summary score | From baseline to weeks 4 and 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on QoL.
  KCCQ overall summary score (no unit, ranges from 0 to 100 with higher scores reflecting better health status).
Proportion of participants with a ≥5, ≥10 and ≥15 point increase in KCCQ clinical and overall summary scores | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on QoL.
  KCCQ clinical summary score (no unit, ranges from 0 to 100 with higher scores reflecting better health status).
  KCCQ overall summary score (no unit, ranges from 0 to 100 with higher scores reflecting better health status).
Change in Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) and Change (DTSQc) | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on QoL.
  Treatment satisfaction status score (no unit, ranges from 0 to 36, with higher scores reflecting greater treatment satisfaction).
  Treatment satisfaction change score (no unit, designed to overcome ceiling effects and to detect changes in treatment satisfaction on a scale from -18 to 18 with negative scores reflecting decreased treatment satisfaction, 0 reflecting no change and positive scores reflecting increased treatment satisfaction).
Change in EQ-5D-5L questionnaire score | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on QoL.
  The instrument consists of two components: the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ-VAS).The first part consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five response levels (level 1 "no problems", level 2 "slight problems", level 3 "moderate problems", level 4 "severe problems", and level 5 "extreme problems"), from which a single EQ-5D index score can be calculated ranging from 0 to 1 where higher scores indicate higher health utility. The EQ-VAS measures one's self-perceived health today on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health) on which participants have to indicate their current health.
Change in distance covered during 6-minute walk test | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on walking distance
Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on NT-proBNP
Change in Haemoglobin A1c (HbA1c) | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on glycaemic control
Proportion of participants with level 2 or level 3 hypoglycaemia | From baseline to weeks 16 and 20
  To provide information on safety and tolerability of sotagliflozin 200mg once daily in addition to standard of care compared to placebo
Proportion of participants with diabetic ketoacidosis (DKA) | From baseline to weeks 16 and 20
  To provide information on safety and tolerability of sotagliflozin 200mg once daily in addition to standard of care compared to placebo
Proportion of participants requiring hospitalisation due to heart failure (HF) | From baseline to weeks 16 and 20
  To provide information on safety and tolerability of sotagliflozin 200mg once daily in addition to standard of care compared to placebo

OTHER OUTCOMES:
Change in New York Heart Association (NYHA) class | From baseline to weeks 16 and 20
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on HF symptoms, signs and clinical outcomes
Change in daily loop diuretic dose | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on HF symptoms, signs and clinical outcomes
Change in systolic and diastolic blood pressure. | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on HF symptoms, signs and clinical outcomes
Number of hospitalizations and deaths (first and total number) due to heart failure | From baseline to weeks 16 and 20
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on HF symptoms, signs and clinical outcomes
Change in estimated glomerular filtration rate (eGFR) | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on renal parameters
Change in serum creatinine | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on renal parameters
Change in urine albumin to creatinine ratio | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on renal parameters
Change in total, basal and bolus insulin doses | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on diabetes-related parameters
Change in in body weight | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on diabetes-related parameters
Mean blood glucose level over preceding 14 days | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on Continuous Glucose Monitor (CGM) metrics
Blood glucose percentage time in range (3.9-10.0 mmol/L) over preceding 14 days | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on Continuous Glucose Monitor (CGM) metrics
Blood glucose percentage time below range (3.0-3.8 mmol/L and <3.0 mmol/L) over preceding 14 days | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on Continuous Glucose Monitor (CGM) metrics
Blood glucose percentage time above range (10.1-13.9mmol/L and >13.9 mmol/L) over preceding 14 days | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on Continuous Glucose Monitor (CGM) metrics
Glycaemic variability index | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on Continuous Glucose Monitor (CGM) metrics
C-peptide level | At baseline
  To investigate if trial outcomes are associated with baseline c-peptide levels
Proportion of participants with non-acidotic ketosis | From baseline to week 16
  To investigate the effect of sotagliflozin 200mg once daily in addition to standard of care on ketone levels

CONTACTS AND LOCATIONS:
Overall Officials: Ify Mordi, MBChB, MD, Principal Investigator — University of Dundee
Locations (15):
- United Kingdom (15):
  - Aberdeen Royal Infirmary, Aberdeen
  - Addenbrookes Hospital, Cambridge
  - Ninewells Hospital, Dundee
  - Royal Infirmary of Edinburgh, Edinburgh
  - Glasgow Royal Infirmary, Glasgow Clinical Research Facility, Glasgow
  - Leicester General Hospital, Leicester
  - Aintree University Hospital, Liverpool
  - Prince Philip Hospital, Llanelli
  - Guy's Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Manchester Royal Infirmary Hospital, Manchester
  - Wythenshawe Hospital, Manchester
  - North Manchester General Hospital, Manchester
  - Northern General Hospital, Sheffield
  - Moorgreen Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Datasets of pseudo-anonymised IPD generated/analysed during the current study will be available upon request from the Chief Investigator (CI) Dr Ify Mordi (i.mordi@dundee.ac.uk) at the end of the trial (i.e. when all endpoints/outcomes have been met, key analyses are complete and results published in peer-reviewed scientific journals). Data will remain available for at least 25 years.
  Data will only be released for legitimate secondary research purposes, where the CI agrees that the proposed use has scientific value and will be carried out to a high standard (in terms of scientific rigour, information governance and security), and that there are resources available to satisfy the request.
  Data will only be released in line with participants' consent, all applicable laws relating to data protection and confidentiality, and any existing contractual obligations. No individual participant data will be released before an appropriate agreement is in place setting out the conditions of release. The agreement will govern data retention, usually stipulating that data recipients must delete their copy of the released data at the end of the planned project.